CLINICAL TRIAL: NCT04771195
Title: Social Factors in the Mental Health of Young Adults: Bridging Psychological and Network Analysis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jamil Zaki, Associate Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 24593; R01MH125974 (NIH)
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Anxiety; Depression; Loneliness; Stress
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Class of 2023 and 2024 (Experimental): Stanford undergraduate students who are expected to graduate in Spring of 2023 or 2024
  Interventions: Behavioral: Examination of students' naturally occurring social ties

INTERVENTIONS:
Behavioral: Examination of students' naturally occurring social ties — In this observational study, features of students' social lives, such as the number of quality of relationships they form, and their subjective loneliness, will be used to predict their mental health and well being at later time points.

SUMMARY:
The central goal of this project is to produce a novel, precise, and comprehensive account of social factors in young adult mental health - using a novel combination of network nominations, ecological momentary assessment, and neuroimaging methods. To that end, the investigators will collect data from two successive classes of college undergraduates (i.e., classes of 2023 and 2024) over the course of their collegiate tenure.

DETAILED DESCRIPTION:
The proposed work will consist of four key components. The investigators will collect data from the class of 2023 in each of their remaining years at college, producing (i) longitudinal data that will allow them to probe the long-term mental health effects of connections made during the transition to college, as well as mental health issues and resilience in the wake of the COVID-19 pandemic as a function of social connectedness. The investigators will leverage this rich dataset to build (ii) prospective quantitative models to predict mental health outcomes later in college based on a range of social factors measured early in college. They will further collect (iii) a longitudinal replication cohort, the class of 2024, allowing to establish the robustness of their initial findings across samples. Finally, the investigators will add (iv) a neuroimaging component to this dataset in a subset of the class of 2024. This will allow them to examine brain "markers" of connectedness, and add them to a prospective model, providing a novel integration across brain, behavior, and community levels of analysis, and a synthetic assessment of social factors in long-term mental health.

ELIGIBILITY:
Inclusion Criteria: Stanford undergraduate students in the classes of 2023 and 2024, as well as all students who reside in their dorms.

-

Exclusion Criteria: People under the age of 18

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Depression | September 2021 - May 2024
  Score on self-reported depression measure: Center for Epidemiological Studies Scale - 10 item version. Range = 0 to 30. Higher scores indicate more depressive symptoms
Anxiety | September 2021 - May 2024
  Score on self-reported anxiety measure: State-Trait Anxiety Inventory - 20 item version. Range = 20 to 80. Higher scores indicate more symptoms of anxiety.

SECONDARY OUTCOMES:
Loneliness | September 2021 - May 2024
  Score on self-reported loneliness measure: University of California Loneliness Scale - 8 item version. Range = 1 to 5. Higher score indicate greater feeling of loneliness.
Stress | September 2021 - May 2024
  Score on self-reported stress measure: Perceived Stress Scale. Range = 1 to 3. Higher scores indicate greater feeling of stress.

CONTACTS AND LOCATIONS:
Overall Officials: Jamil Zaki, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Unidentifiable data will be shared with other researchers. To that end, alphanumeric identifiers will be assigned to each individual in the sample's population. Direct nomination lists will not be shared because the potential traceability for participants who may gain access to the data after it is published.
Supporting Information: Study Protocol, SAP, Analytic Code